CLINICAL TRIAL: NCT00887497
Title: Ischemic Conditioning (Delay Phenomenon) in Colorectal Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: terminated due to failure to enroll patients after two years of approval
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-6618
Record Dates: First submitted 2009-04-22; First posted 2009-04-24 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Colon Rectal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Catheterization (Experimental): Patients receive angioembolization prior to surgery
  Interventions: Procedure: Angioembolization

INTERVENTIONS:
Procedure: Angioembolization — Angioembolization

SUMMARY:
One of the major complications of surgical excision of colorectal cancer includes improper healing of the anastomosis (reconnection of the remaining, cancer free intestine). This can result in anastomotic leak, abscess then abdominal and/or pelvic sepsis and mortality.

Esophageal surgery has suffered from complications. Recently, an innovation in esophageal surgery has seen a relatively drastic decrease in complications during distal esophagectomies using a technique called "ischemic conditioning". This technique involves dividing the blood supply to the stomach that would be performed during a 1-stage esophagectomy but returning days later to complete the resection. Bench results have shown improved angiogenesis, vasodilation, less anastomotic collagen deposition and minimized ischemia at the time of surgery while clinical results have included improved stricture rates, leak rates and mortality in esophageal surgery.

Hypothesis Ischemic conditioning is universal to the intestinal tract and a similar technique can be applied in colon and rectal surgery. The investigators plan evaluating this hypothesis by performing a pilot study comprised of the following: performing an endovascular embolization of the inferior mesenteric artery (IMA) followed by interval laparoscopic or open rectosigmoid resection.

Methods Part 1 - Endovascular Procedure Patients will be admitted and undergo endovascular embolization of their IMA as an outpatient following diagnostic angiography. They will undergo sigmoidoscopy throughout the embolization and a laser probe will indirectly measure tissue oxygenation. The patient will be released home that day.

Part 2 - Colorectal Procedure Patients will then return 2-4 days later for their definitive laparoscopic or open rectosigmoid resection. They will undergo sigmoidoscopy before and after surgery and a laser probe will indirectly measure tissue oxygenation. The patient will then be released home on average 3-5 days later.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety and feasibility of ischemic conditioning of the colon prior to resection. Colon and rectal resections require the removal of a section of colon or rectum with re-attachment (anastomosis) of the two ends. This joining together of the intestine is at risk for leaking if healing does not occur appropriately. Factors postulated to lead to anastomotic leak include ischemia as well as tension and infection among others.

The concept of ischemic conditioning is based upon the innate ability to compensate and increase the blood flow to a section of the intestine which is locally ischemic. By inducing ischemia to a segment of intestine prior to resection, one could theoretically increase blood flow via collateral vessels prior to resection. This would then, in turn, lead to more initial blood flow to an anastomosis at the time of surgery via these collaterals, thereby decreasing ischemia to a new, healing anastomosis.

Ischemic conditioning was first described in animal models proving its safety and efficacy. In the rat model, ischemic conditioning demonstrated a return to baseline of tissue perfusion by the time of resection, improved anastomotic leak rate and higher anastomotic wound breaking strength. The first time this idea was implemented in the human model was in a study by Akiyama et. al. where preoperative embolization was shown to be safe and improved blood supply to the distal end of anastomosis after esophagectomy (remaining stomach). Further basic science studies have shown improved angiogenesis, vasodilation, less anastomotic collagen deposition and minimized ischemic injury. Further clinical studies demonstrated improved stricture rates (0% from 40%), leak rates (0-6% from 5-15%) and mortality (0% from 5-10%).

One of the major complications in colon and rectal surgery is improper healing of the anastomosis (connection between the remaining, cancer free rectum with the remaining colon). This results in an anastomotic leak or dehiscence leading to abscess, abdominal sepsis requiring longer hospital stays, IV antibiotics, reoperation or possibly even death. It can also lead to the late complication of stricture impairing function and often requiring repeat dilations or operative revision. Recent reviews show rates of anastomotic complications in upper rectal resection at 8-17% for leaks, and an average hospital stay of 10 days.

In the current study, preoperative embolization of the Inferior Mesenteric Artery (IMA) is performed for patients scheduled to undergo colon or rectal resection. The surgery is then performed in the standard fashion (either laparoscopically or open) several days later (1-5 days). The study is designed as a prospective, non-randomized, safety (pilot) study. Since there are no reports of performing this exact procedure, we feel it is necessary to initially proceed with safety study without a comparative arm prior to a large scale, multicenter trial evaluating outcomes. Therefore, in this study we will not be evaluating morbidity or mortality outcomes to any statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age, male or female
* Are scheduled for a non-emergent, resection of your colon
* Are able to give written informed consent to indicate an understanding of the study procedures.

Exclusion Criteria

* Will be undergoing an emergency procedure or has a diagnosis of bowel complication(s) such as bowel obstruction, constriction, inflammation, infection, or have inflammatory bowel disease.
* Are currently participating in another clinical trial which may affect this study's outcomes.
* Have been taking regular steroid medication.
* Have a negative reaction to general anesthesia.
* Have severe arterial occlusive disease (disease of the blood vessels affecting blood flow to your legs).
* Have an abdominal aortic aneurysm (dilation of the large artery in your abdomen).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Any adverse even (safety study) | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Mills, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States